CLINICAL TRIAL: NCT02223416
Title: A Study Aimed at Assessing the Pharmacokinetic Properties of RGB-10 and Forsteo
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Gedeon Richter Plc. (Industry)
Responsible Party: Sponsor
Other Study IDs: RGB-10-001
Record Dates: First submitted 2014-08-21; First posted 2014-08-22 (Estimated); Last update posted 2015-03-18 (Estimated); Status verified 2014-08

CONDITIONS: Healthy
Keywords: female; volunteers
MeSH Terms: interventions — RGB-10; Teriparatide

ARMS (2):
- RGB-10 (Experimental)
  Interventions: Drug: RGB-10
- Forsteo (Active Comparator)
  Interventions: Drug: Teriparatide

INTERVENTIONS:
Drug: RGB-10
  Arms: RGB-10
Drug: Teriparatide
  Arms: Forsteo

SUMMARY:
Pharmacokinetic properties, safety and tolerability of RGB-10 and Forsteo will be compared in healthy female volunteers.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adult female subjects
* 18-55 years of age (inclusive)
* BMI must be between 18.5 and 27 kg/m2 (inclusive)

Exclusion Criteria:

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Dates: Primary Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
Area under the plasma concentration versus time curve (AUC) | 0-4 hours
Peak Plasma Concentration (Cmax) | 0-4 hours

CONTACTS AND LOCATIONS:
Locations (1):
- Celerion (UK), Belfast, United Kingdom